CLINICAL TRIAL: NCT01856374
Title: Serial EValuation of multiplE Coronary Artery Diseases by an Optical Coherence Tomography; Assessment of the Changes of de Novo Lesions and Comparisons of Neointimal Coverage Between Xience Prime® Versus Cypher SelectTM Stents; SEVEN-Xience Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2010-0052
Record Dates: First submitted 2013-05-09; First posted 2013-05-17 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Multi-vessel Diseases, Angina
MeSH Terms: conditions — Angina Pectoris | interventions — Pravastatin; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cypher group (Active Comparator)
  Interventions: Device: Sirolimus-eluting stent (Cypher SelectTM, Cordis, Miami, FL)
- Xience group (Experimental)
  Interventions: Device: Everolimus-eluting stent(Xience Prime®, Abbott Vascular, Santa Claea, CA)
- Pravastatin group (Active Comparator)
  Interventions: Drug: Pravastatin 20mg
- Atorvastatin group (Experimental)
  Interventions: Drug: Atorvastatin 40mg

INTERVENTIONS:
Device: Sirolimus-eluting stent (Cypher SelectTM, Cordis, Miami, FL) — Patients with native coronary arteries fulfilling all enrollment criteria will be randomly assigned to each DES group; Xience Prime® vs. Cypher SelectTM and pravastatin 20mg vs. atorvastatin 40mg.
  Arms: Cypher group
Device: Everolimus-eluting stent(Xience Prime®, Abbott Vascular, Santa Claea, CA) — Patients with native coronary arteries fulfilling all enrollment criteria will be randomly assigned to each DES group; Xience Prime® vs. Cypher SelectTM and pravastatin 20mg vs. atorvastatin 40mg.
  Arms: Xience group
Drug: Pravastatin 20mg — 2x2 randomization by the treatment of dyslipidemia (In patients of dyslipidemia: pravastatin 20mg/day vs. atorvastatin 40mg and the types of the implanted cypher vs xience.
  Arms: Pravastatin group
Drug: Atorvastatin 40mg — 2x2 randomization by the treatment of dyslipidemia (In patients of dyslipidemia: pravastatin 20mg/day vs. atorvastatin 40mg and the types of the implanted cypher vs xience.
  Arms: Atorvastatin group

SUMMARY:
This study is a prospective open-labeled, randomized study to compare the neointimal coverage at 3 months and 12 months and its serial changes between 3 months and 12 months according to the implanted DES and evaluate the serial changes in the proximal portions of 3 epicardial coronary artery and left main artery including the assessment of fibrous cap thickness and lipid pool for vulnerable plaques by OCT. In addition, the investigators will compare the changes such as plaques and neointimal coverage from serial OCT follow-up according to the different statin strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 20 years old
* Patients with typical angina who are considered for coronary revascularization.
* Multi-vessel diseases: more than 2 significant coronary de novo lesions (> 70% by quantitative angiographic analysis); one of the target lesions is the most significant tight stenotic lesion causing the ischemic symptom and requiring the immediate revascularization but the others are significant but non-tight lesions to be delayed or observed for 3 months and not requiring immediate PCI for the complete revascularization of all coronary arteries.

Exclusion Criteria:

* ST-elevation MI
* Cardiogenic shock or hemodynamically unstable status
* Lesions requiring the immediate complete revascularization of all coronary stenotic lesions
* Contraindication to anti-platelet agents
* Treated with any DES within 6 months at other vessel
* Creatinine level ≥ 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Pregnant women or women with potential childbearing
* Life expectancy 1 year
* Complex lesion morphologies (bifurcation lesions treated with 2-stent techniques, untreated significant unprotected left main diseases, chronic total occlusion, in-stent restenosis, and vein graft lesion)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
neointimal coverage according to the implanted DES; Xience vs. Cypher | up to 12month after stent implantation
  Neointimal coverage means percentage of uncovered struts on OCT. The percentages of uncovered struts were compared between EES and SES.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim JS, Kim JH, Shin DH, Kim BK, Ko YG, Choi D, Jang Y, Hong MK. Effect of High-Dose Statin Therapy on Drug-Eluting Stent Strut Coverage. Arterioscler Thromb Vasc Biol. 2015 Nov;35(11):2460-7. doi: 10.1161/ATVBAHA.115.306037. Epub 2015 Sep 10. PMID 26359512